CLINICAL TRIAL: NCT02178059
Title: An Open-label, Single-dose, 2-period Cross Over Study in Healthy Volunteers to Assess Relative Bioavailability of Terbutaline Sulphate 1.5 mg After Inhalation Via the M3 Turbuhaler Compared With the M2 Turbuhaler
Brief Title: Relative Bioavailability Study to Compare Inhalation of Terbutaline Sulphate 1,5mg Via Turbuhaler M3 With Turbuhaler M2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4711C00002
Record Dates: First submitted 2014-06-27; First posted 2014-06-30 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers, pharmacokinetic, inhalation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bricanyl Turbuhaler M3 (Experimental): 0.4 mg terbutaline sulphate (delivered dose) per inhalation
  Interventions: Drug: terbutaline sulphate delivered dose
- Bricanyl Turbuhaler M2 (Active Comparator): 0.5 mg terbutaline sulphate (metered dose) per inhalation
  Interventions: Drug: terbutaline sulphate metered dose

INTERVENTIONS:
Drug: terbutaline sulphate delivered dose — 0.4 mg terbutaline sulphate (delivered dose) per inhalation
  Other Names: Turbuhaler New Version
  Arms: Bricanyl Turbuhaler M3
Drug: terbutaline sulphate metered dose — 0.5 mg terbutaline sulphate (metered dose) per inhalation
  Other Names: Turbuhaler Current Version
  Arms: Bricanyl Turbuhaler M2

SUMMARY:
Relative bioavailability study to compare inhalation of Terbutaline Sulphate 1,5mg via current version of Turbuhaler with inhalation via a new version

DETAILED DESCRIPTION:
An Open-label, Single-dose, 2-period Cross over Study in Healthy Male and Female Volunteers to Assess Relative Bioavailability of Terbutaline Sulphate 1.5 mg after Inhalation via the M3 Turbuhaler (New Version) Compared with the M2 Turbuhaler (Current Version)

ELIGIBILITY:
Inclusion Criteria:

1. Female and male volunteers aged between 18 and 65 years, both inclusive
2. Healthy as judged by the Principal Investigator after medical history, physical examination, 12-lead ECG, laboratory tests (including HIV, HBsAg and hepatitis C antibody tests) and assessments of pulse rate and blood pressure
3. Ability to use a Turbuhaler according to the provided instructions, as judged by the Principal Investigator or the study nurse
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weighing at least 50 kg and no more than 100 kg -

Exclusion Criteria:

1. History or presence of respiratory, gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs (except for cholecystectomy)
2. Current smokers or those who have smoked or used nicotine products within the previous 3 months should be excluded
3. Plasma donation within 1 month of screening or any blood donation or blood loss of more than 500 mL during the 3 months prior to screening
4. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Principal Investigator or history of hypersensitivity to terbutaline (or drugs of a similar chemical structure or class) or inhaled lactose
5. Positive screen for drugs of abuse and/or alcohol and/or cotinine at screening (Visit 1) or on admission to the study centre (Day -1) prior to administration of the investigational medical product (IMP) on Day 1 -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amitava Ganguli, MB ChB, MRCP, Principal Investigator — Quintiles London United Kingdom; Göran Eckervall, MD, Study Director — Astrazeneca Mölndal, Sweden; Ola Beckman, MD, Study Chair — Astrazeneca Mölndal, Sweden
Locations (1):
- Research Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single centre study conducted in the UK.
Pre-assignment Details: Healthy subjects were assessed for eligibility at a screening visit (Visit 1) within 28 days of administration of the first dose of terbutaline via Bricanyl Turbuhaler M2 or Bricanyl Turbuhaler M3 (Visit 2). Subjects were randomly assigned to 1 of 2 treatment sequences: M3 then M2 or M2 then M3
Groups:
- M3 First, Then M2: Sequence 1: M3 first then M2
- M2 First, Then M3: Sequence 2: M2 first, then M3
Period: First Intervention
Arm/Group | M3 First, Then M2 | M2 First, Then M3
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: Washout
Arm/Group | M3 First, Then M2 | M2 First, Then M3
Started | 17 | 17
Completed | 16 | 17
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Second Intervention
Arm/Group | M3 First, Then M2 | M2 First, Then M3
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects
Groups:
- Randomized Subjects: All randomized subjects
Arm/Group | Randomized Subjects
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11)
Gender [Count of Participants; unit: Participants]
  Female | 18
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Zero to the Time of Last Measurable Concentration [AUC(0-t)]
Description: These will be taken at each treatment period
Time Frame: Samples will be taken at predose, and at 5, 10, 20, 40, 80, 100 minutes and at 2, 4, 6, 9, 12, 18, 24, 30, and 36 hours postdose
Population: The PK analysis set included all healthy subjects who received at least 1 dose of the IMP and had at least 1 postdose PK measurement without important protocol deviations/violations or events thought to significantly affect the PK of the IMP.
Measure: Geometric Mean (95% Confidence Interval); unit: nmol*h/L
Groups:
- Bricanyl Turbuhaler M3: Bricanyl Turbuhaler M3: 0.4 mg terbutaline sulphate (delivered dose) per inhalation
- Bricanyl Turbuhaler M2: Bricanyl Turbuhaler M2: 0.5 mg terbutaline sulphate (metered dose) per inhalation
Arm/Group | Bricanyl Turbuhaler M3 | Bricanyl Turbuhaler M2
Number analyzed (Participants) | 34 | 33
nmol*h/L | 89.04 [80.84 to 98.07] | 100.9 [91.54 to 111.3]
Statistical Analysis 1: Comparison: Bricanyl Turbuhaler M3 vs Bricanyl Turbuhaler M2; No increase in the exposure of plasma terbutaline after administration of Bricanyl Turbuhaler M3 will be concluded if the upper bound of the 90% CIs for the ratios of AUC and Cmax are both below 1.25; Test type: Non-Inferiority or Equivalence — Approximately 34 healthy volunteers will be entered into the study in order to complete 30 evaluable volunteers. Based on the study SD-001-0268, a residual intra-individual standard deviation of 0.300/sqrt(2) = 0.212 can be expected on the natural log scale. With 30 completed volunteers there will be a 93% chance that the upper limits of two-sided 90% CI for Cmax and AUC ratios are <1.25 provided that the true mean ratios are <1.05; Ratio of geometric means (%) = 88.20, 90% CI 2-sided [81.03 to 96.02] — Comparison of Bricanyl Turbuhaler M3 (test) to Bricanyl Turbuhaler M2 (reference)

2. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: These will be taken at each treatment period
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hour
Arm/Group | Bricanyl Turbuhaler M3 | Bricanyl Turbuhaler M2
Number analyzed (Participants) | 34 | 33
hour | 1.33 [1.33 to 1.67] | 1.33 [1.33 to 1.67]
Statistical Analysis 1: Comparison: Bricanyl Turbuhaler M3 vs Bricanyl Turbuhaler M2; Test type: Superiority or Other; p = 0.8052, Wilcoxon signed rank test; Median Difference (Final Values) = 0.00, 90% CI 2-sided [-0.17 to 0.17]

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero Extrapolated to Infinity (AUC)
Description: These will be taken at each treatment period
Time Frame: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol*h/L
Arm/Group | Bricanyl Turbuhaler M3 | Bricanyl Turbuhaler M2
Number analyzed (Participants) | 34 | 33
nmol*h/L | 96.63 [87.68 to 106.5] | 109.7 [99.43 to 121.0]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to 36 Hours Postdose [AUC(0-36)]
Description: These will be taken at each treatment period
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Bricanyl Turbuhaler M3 | Bricanyl Turbuhaler M2
Number analyzed (Participants) | 34 | 33
nmol*h/L | 89.0 (29.5) | 101 (27.8)

5. Secondary Outcome: Terminal Half-life (t1/2)
Description: These will be taken at each treatment period
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Bricanyl Turbuhaler M3 | Bricanyl Turbuhaler M2
Number analyzed (Participants) | 34 | 33
hour | 11.7 (8.9) | 11.8 (10.9)

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: These will be taken at each treatment period
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Bricanyl Turbuhaler M3 | Bricanyl Turbuhaler M2
Number analyzed (Participants) | 34 | 33
nmol/L | 12.00 [10.73 to 13.40] | 13.12 [11.73 to 14.67]
Statistical Analysis 1: Comparison: Bricanyl Turbuhaler M3 vs Bricanyl Turbuhaler M2; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric means (%) = 91.44, 90% CI 2-sided [84.82 to 98.58] — Comparison of Bricanyl Turbuhaler M3 (test) to Bricanyl Turbuhaler M2 (reference)

ADVERSE EVENTS:
Arm/Group | Bricanyl Turbuhaler M3 | Bricanyl Turbuhaler M2
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 12/34 | 11/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bricanyl Turbuhaler M3 (N=34) | Bricanyl Turbuhaler M2 (N=33)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 9 (10) | 7 (8)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.